CLINICAL TRIAL: NCT00379054
Title: Intervention for Support Persons to Help Smokers Quit
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1928-04; 5R21DA018365-02 (NIH); 1R21DA018365-01 (NIH)
Record Dates: First submitted 2006-09-19; First posted 2006-09-21 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2010-11

CONDITIONS: Smoking Cessation
Keywords: social support, smoking, smoking cessation, intervention,; telephone counseling
MeSH Terms: conditions — Smoking Cessation; Smoking

INTERVENTIONS:
Behavioral: telephone based skills training intervention

SUMMARY:
This study will examine the feasibility and potential effectiveness of an intervention for adults who want to help support a smoker to quit. The support persons will receive either self-help materials only or the self-help materials plus a telephone counseling intervention. Both interventions provide information on how support persons can encourage a smoker to quit.

DETAILED DESCRIPTION:
Interventions that reach the majority of cigarette smokers in the population have the greatest potential to impact the public health. Most smokers do not seek treatment for smoking cessation. A novel behavioral approach to reaching smokers is to directly recruit and train adult nonsmokers to intervene (i.e., support persons). Several studies provide evidence for the role of social support in smoking cessation. The use of support persons as change agents for smoking cessation represents a shift from conventional interventions that focus almost exclusively on the smoker. This proposal builds on our previous work that indicates a skills training intervention for support persons is feasible and acceptable to participants. Moreover, the effect size observed for the smoking abstinence rate in the smokers, as reported by the support persons, provides some evidence of potential efficacy. However, the intensive, group, clinic-based format of the intervention limits its potential dissemination. We propose to develop and pilot test a more streamlined version of the intervention using a telephone-based format. To enhance internal validity of the findings, additional formative work is also needed to examine the feasibility of obtaining baseline assessments and outcomes directly from the smoker. Social cognitive theory is the conceptual basis for the proposed intervention.

The objective of this R21 proposal is to develop and pilot test a novel behavioral approach to smoking cessation that utilizes support persons in the smoker's natural environment. We expect that as a result of this project, we will have developed a well-specified and feasible telephone counseling intervention, the efficacy of which can be tested in future larger-scale randomized clinical trials.

This project will take place in two phases. In Phase 1, we will develop a telephone counseling intervention for support persons, adapting and refining the intervention from our previous, clinic-based treatment study. During this phase, we will develop the telephone counselor manual, and 10 support persons will complete the protocol, which will be modified and refined based on feedback from participants and counselors. Phase 2, consisting of a pilot clinical trial, will apply a randomized, two group design with repeated assessments at weeks 0 (baseline), 10 (end-of-treatment), and 26. Support persons (N=60) will be recruited and randomly assigned to self-help intervention or telephone counseling. The smokers will be enrolled as study subjects but will be contacted for assessments only.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, the support person must (1) be 18 years of age or older, (2) provide written informed consent, (3) be a never or former cigarette smoker (no cigarette use during the past 6 months), (4) be interested in helping someone 18 years of age who is a current smoker (average of 10 cigarettes per day in the past 7 days), (5) be able and willing to participate in all aspects of the study, (6) have current and anticipated contact (any combination of face-to-face, telephone, or electronic mail) with the smoker a total of at least 4 days of the week for the study duration, and (7), the smoker provides informed consent for the support person's involvement in the study.

-

Exclusion Criteria:

(1) another support person from the same household has enrolled, (2) another support person has enrolled to help the same smoker, or (3) the smoker is currently (past 30 days) receiving pharmacologic or behavioral treatment for nicotine dependence.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2005-09; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Feasibility (recruitment and retention of support persons and smokers),
acceptability of intervention to support persons, potential efficacy
(determined by number of smoker quit attempts, smoking abstinence, readiness
to quit)and changes in supportive behaviors among the support persons as
measured by the Support Provided Measure.

CONTACTS AND LOCATIONS:
Overall Officials: Christi A Patten, Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo, Rochester, Minnesota, United States